CLINICAL TRIAL: NCT05402124
Title: The Colorectal Cancer Chemoprevention Acceleration and Improvement Platform (CRC-CHAMP) Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CRC-CHAMP01
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colorectal Adenomatous Polyp
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, prospective cohort pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASA 81mg (Other): Acetylsalicylic acid delayed release tablets (81mg), single tablet taken once per day for 90 days.
  Interventions: Drug: acetylsalicylic acid delayed release tablets, 81mg

INTERVENTIONS:
Drug: acetylsalicylic acid delayed release tablets, 81mg — acetylsalicylic acid delayed release tablets, 81mg taken once per day for 90 days
  Other Names: ASPIRIN 81mg; Drug Identification Number 02237726

SUMMARY:
The overall goal of this study is to develop a platform for both large-scale chemoprevention trials and real-world chemoprevention studies for colorectal cancer (CRC) prevention. The specific objectives of this proof of concept study are to:

1. Evaluate the feasibility of a real-world chemoprevention agent (CPA) intervention (3-months of daily low-dose acetylsalicylic (ASA)) in participants at increased risk for CRC (one or more high-risk adenomas removed during colonoscopy) based on participant uptake, adherence (days taking CPA), and adverse events;
2. Evaluate factors related to uptake and adherence of ASA using validated surveys and interviews.

DETAILED DESCRIPTION:
Study Design and Duration:

This is a single arm (non-randomized), open-label prospective cohort pilot study.

Screening Phase: up to 2 weeks Treatment Phase: 90 days Follow-up Phase: 90 days

Screening Phase: up to 14 days. Participants will consent to being enrolled in the study and to the use of ASA for a 90 day period. Regardless of agreement to use ASA for the entire study period, all participants will complete 6 baseline questionnaires.

Active Treatment Phase: up to 90 days. Participants that agree to the use of ASAs will be instructed to take daily ASAs for 90 days. Participants will be contacted by telephone at 1, 2, and 3 months to determine adverse events, adherence, and discontinuation. At 3 months participants will fill out a chemoprevention questionnaire and the Adherence Barriers Questionnaire (ABQ).

Follow-up Phase: 90 days. During the follow-up phase, participants will not be provided with ASA through the study nor will a specific recommendation be made to continue ASA. All participants will be contacted via telephone at the end of this period to determine the prevalence of continued use of ASA on their own.

Total study commitment will be up to 194 days. After consent, participants complete a 90 day active treatment phase followed by a 90 day follow-up phase. The trial is expected to be completed within one year.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 50-59 at time of signing the informed consent
2. Documented history of high-risk adenomatous polyps diagnosed within the previous 12 months:

   1. At least one villous or tubulovillous polyp of any size
   2. At least one polyp with high-grade dysplasia of any size
   3. At least one adenomatous polyp ≥1 cm in size
   4. Three or more tubular adenomas <1 cm in size
3. Not currently using ASA for another condition

Exclusion Criteria:

1. Age < 50 or >= 60
2. Known allergy or hypersensitivity to ASA, salicylates or non-steroidal anti- inflammatory drugs.
3. Daily alcohol use > 3 units
4. Regular use of aspirin or non-steroidal anti-inflammatory drugs (> 2 dose/week)
5. Current use of corticosteroid (any dose) orally
6. Current use of methotrexate, valproic acid or digoxin
7. Currently taking any anti-cancer drug
8. Current use of anti-platelet agents or anticoagulants
9. Anticipated surgical procedure in the next 3 months
10. Current or past history of gastrointestinal ulcers
11. History of gastrointestinal bleeding (except hemorrhoidal or minor outlet type bleeding)
12. Known cirrhosis or hepatic impairment (for example, total bilirubin >1.25 Upper Limit of Normal, International Normalized Ratio >1.25)
13. Known bleeding disorder (hemorrhagic diathesis)
14. History of asthma or nasal polyps
15. History of colorectal cancer
16. Platelet count < 120 or > 450 (within previous 3 months)
17. Renal insufficiency (eGFR < 90 within previous 3 months)
18. History of congestive heart failure or left ventricular ejection fraction < 50 percent

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Uptake of ASA | 7 days
  Initiation of daily ASA 81mg (Percentage of participants who complete first 7 days of treatment).
Adherence to ASA over 90 days | 90 days
  Number of days taking ASA over a 90 day period. The time (number of days) on ASA for participants that discontinued use will be quantified.
Adherence to at least 50 percent of total prescribed dose | 90 days
  Percentage of participants who take at least 50 percent of total prescribed dose. Descriptive statistics will be utilized to characterize participants that adhered to ASA and participants who did not.
Measurement of Adverse Events | 90 days
  Measurement of Adverse Events reported through interviews with research study nurse and participant report over 90 days (active treatment phase).

SECONDARY OUTCOMES:
Factors related to uptake and adherence to ASA | From enrollment to 90 days
  Behavioral, sociodemographic and health characteristics, measured using Health & Lifestyle Questionnaire and presented as percentages.
Factors related to uptake and adherence to ASA using measurement of health related quality of life | At enrollment
  Behavioral, sociodemographic and health characteristics, measured using Short-Form 36 Health Survey Questionnaire to measure quality of life and presented as percentages.
Factors related to uptake and adherence to ASA using measurement of self efficacy | At enrollment
  Behavioral, sociodemographic and health characteristics, measured using National Institutes of Health (NIH) Self-efficacy questionnaire and presented as percentages.
Factors related to uptake and adherence to ASA | At enrollment
  Measurement of beliefs, attitudes and values about medicines using Beliefs about Medicines questionnaire and expressed as percentages.
Factors related to uptake, in-study adherence and post-study maintenance using measurement of adherence barriers | At enrollment through end of treatment at 90 days
  Measurement of Adherence barriers using Adherence Barriers Questionnaire (at baseline and 3m follow-up) and expressed as percentages.
Factors related to uptake, in-study adherence and post-study maintenance using measurement of chemoprevention knowledge | At enrollment through end of treatment at 90 days
  Measurement of knowledge about chemoprevention using Chemoprevention Questionnaires (baseline and 3m follow-up) and expressed as percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hilsden, Principal Investigator — University of Calgary
Locations (1):
- Forzani & Macphail Colon Cancer Screening Centre, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers other than the Principal and Co-investigators. The results of this study will be published in a scientific peer reviewed journal. Both the chemoprevention intervention results and the feasibility results for scaling a chemoprevention program to all individuals attending a screening center will be presented. The qualified investigator holds the primary responsibility for publication of study results.